CLINICAL TRIAL: NCT03778853
Title: An Open, Single-arm, Multi-center Study of Anlotinib in Advanced Non-squamous NSCLC Patients in the Elderly Without Systemic Chemotherapy
Brief Title: Study of Anlotinib in Advanced Non-squamous NSCLC Patients in the Elderly Without Systemic Chemotherapy (ALTER-L006)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: LanZhou University (Other)
Collaborators: General Hospital of Ningxia Medical University (Other)
Responsible Party: Principal Investigator, Chen Rui, professor, LanZhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20180049
Record Dates: First submitted 2018-12-15; First posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Advanced Non-squamous NSCLC
Keywords: Non-squamous NSCLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib Hydrochloride (Experimental): Anlotinib Hydrochloride p.o, qd and it should be continued until disease progress or toxicity cannot be tolerated or patients withdraw consent
  Interventions: Drug: Anlotinib Hydrochloride

INTERVENTIONS:
Drug: Anlotinib Hydrochloride — Anlotinib Hydrochloride ( 12mg, QD, PO, d1-14, 21 days per cycle), take once when limosis in the morning. If patients cannot suffer from AEs, they can get declined dosage.
  Other Name: AL3818

SUMMARY:
Anlotinib is a multi-target receptor tyrosine kinase inhibitor in domestic research and development. It can inhibit the angiogenesis related kinase, such as VEGFR, FGFR, PDGFR, and tumor celltebiz related kinase -c-Kit kinase. In the phase III study, Patients who failed at least two kinds of systemic chemotherapy (third line or beyond) or drug intolerance were treated with anlotinib (12mg, po. qd. on day 1to14 of a 21-day cycle) or placebo, the anlotinib group PFS and OS were 5.37 months and 9.63 months, the placebo group PFS and OS were 1.4 months and 6.3 months.

DETAILED DESCRIPTION:
It is an open, single-arm, multi-center clinical trial conducted in China, and plan to Recruiting 72 patients in the elderly without systemic chemotherapy. Patents receive 12mg anlotinib orally daily on day 1to 14 of a 21-day cycle until progression of disease, assess safety and efficacy of the drug.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent
* Age：≥70
* Subjects with histologically or cytologically confirmed locally advanced and/or advanced NSCLC
* at least two systematic chemotherapy with upwards of 1-line treatments or cannot suffer
* The negative patients in EGFR&ALK can participate or who positive in EGFR&ALK, have or have not drug tolerance after the treatment with relative targeted drugs
* Subjects with at least one measurable lesion as defined by RECIST (version 1.1)
* Expected Survival Time: Over 3 months
* ECOG PS：0-1
* main organs function is normal

Exclusion Criteria:

* 1.Small Cell Lung Cancer (including small cell cancer and other kinds of cancer mixed with non-small cell cancer)
* lung squamous carcinoma
* Other active malignancies requiring treatment
* History of malignancy
* Have got non remissive toxic reactions derived from previous therapies, which is over level 1 in CTC AE (4.0), alopecia NOT included
* Abnormal coagulation (INR>1.5 or PT>ULN+4s or APTT >1.5 ULN); Patients with any physical signs of bleeding diathesis or receiving thrombolysis and anticoagulation
* take major surgical treatments or have serious trauma before grouping, or the impact of surgery or trauma has been eliminated for less than 14 days
* Patients with active or unable to control serious infections
* Patients with Grade II or higher myocardial ischemia, myocardial infarction or malignant arrhythmias(including QTc male ≥ 450 ms, female ≥ 470 ms) ; Patients with grade III to IV cardiac insufficiency, or left ventricular ejection fraction (LVEF) <50% (NYHA Classification)
* Patients with non-healing wounds or fractures
* with kinds of factors which affect oral medicine (e.g. failing to swallow, gastrointestinal tract getting resected, chronic diarrhea and ileus).
* get arterial/venous thrombosis within 12 months, such as cerebrovascular accidents (including temporary ischemic stoke), deevenous thrombosis, and pulmonary embolism
* Patients with cirrhosis, decompensated liver disease, or active hepatitis Have suffered from hemorrhagic disease or coagulation dysfunction
* diagnosed with disease which will severely endanger the security of patients or influence the completion of this research

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
PFS | Time Frame: each 42 days up to PD or death(up to 24 months)
  Progress free survival (PFS)

SECONDARY OUTCOMES:
OS | From randomization until death (up to 24 months)
  Overall Survival (OS)
DCR | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  Disease Control Rate (DCR)
ORR | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  Objective Response Rate (ORR)
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Until 30 day safety follow-up visit
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability
EORTC QLQ-C30 | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  use EORTC QLQ-C30(version 3) questionnaire to evaluate the quality of life

CONTACTS AND LOCATIONS:
Overall Officials: xiaoming hou, professor, Principal Investigator — LanZhou University

IPD SHARING:
Plan to Share IPD: Undecided